CLINICAL TRIAL: NCT06726096
Title: Randomized,Double-blind,Placebo,Positive-controlled Phase III Trial of VDJ001 In Patients With Moderate-to-severe Active Rheumatoid Arthritis
Brief Title: Phase III Trial of VDJ001 In Patients With Moderate-to-severe Active Rheumatoid Arthritis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing VDJBio Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VDJ001-RA-Ⅲ
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA); Anti IL-6R
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combinant humanized monoclonal antibody against interleukin-6 receptor 6 mg/kg (Experimental)
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection
- placebo control (Placebo Comparator)
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection
- Tocilizumab Injection 8 mg/kg (Active Comparator)
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection

INTERVENTIONS:
Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection — The drug was administered once every 4 weeks.
  Other Names:
  Tocilizumab Injection placebo control

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, and active drug-controlled Phase III pivotal clinical trial of recombinant humanized anti-interleukin-6 receptor monoclonal antibody injection (VDJ001) for the treatment of moderate-to-severe active rheumatoid arthritis with poor response to methotrexate

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. Age between 18 and 75 years inclusive;
3. Diagnosed with RA according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 ACR and European League Against Rheumatism (EULAR) classification criteria;
4. At the time of screening, judged to have moderate to severe active RA based on the following criteria: joint swelling count ≥6 (out of 66 joints) and joint tenderness count ≥6 (out of 68 joints), and must also meet C-reactive protein (CRP)/High-sensitivity C-reactive protein (hsCRP) ≥ upper limit of normal (ULN) or erythrocyte sedimentation rate (ESR) ≥28 mm/h;
5. Have been receiving oral methotrexate (MTX) treatment for at least 12 weeks and at a stable dose (MTX dose of 7.5~25 mg/week) for at least 4 weeks prior to randomization; subjects with a history of parenteral MTX (subcutaneous, intramuscular, or intravenous injection) are eligible for the study, but these subjects must have been receiving a stable dose of MTX 7.5~25 mg/week oral treatment for ≥4 weeks prior to randomization;
6. At the time of screening, if the subject is taking prednisone or an equivalent dose of corticosteroids, they must have been on a stable dose (prednisone dose ≤10mg/day) for at least 4 weeks prior to randomization.

Exclusion Criteria:

1. Body weight >100 kg or <40 kg;
2. ACR functional class IV or long-term bedridden/wheelchair-bound individuals;
3. Individuals with an allergic constitution or known allergies to any components of the study treatment or other similar products;
4. Investigators determine that surgeries previously received by the subject or planned surgeries may affect the assessment of joint study evaluations;
5. Patients with rheumatic immune diseases other than rheumatoid arthritis, uncontrolled immune system diseases requiring oral corticosteroid treatment, which the investigator deems may affect trial evaluation;
6. Primary or secondary immunodeficiency diseases (past or currently active);
7. History of or current tumors (except for cured and non-recurrence for at least 5 years of skin basal cell carcinoma, squamous cell carcinoma, cervical carcinoma in situ, breast ductal carcinoma in situ, and papillary thyroid carcinoma);
8. History of any lymphoproliferative diseases, such as EBV-related lymphoproliferative diseases, lymphoma, leukemia, myeloproliferative diseases, multiple myeloma, or signs and symptoms suggesting current lymphatic diseases;
9. Presence of severe, poorly controlled comorbidities, such as (but not limited to) neurological, cardiovascular, liver, kidney, gastrointestinal, endocrine diseases, which the investigator judges may hinder the subject's participation in this study;
10. Known to have the following infections: recurrent active bacterial, viral, fungal, mycobacterial, or other infections [including but not limited to tuberculosis and atypical mycobacterial disease, granulomatous disease found on chest X-ray, hepatitis C virus infection, human immunodeficiency virus (HIV) infection, and herpes zoster, but excluding nail bed fungal infections], or a history of chronic infections within the last 6 months, or any major infection requiring hospitalization for treatment or intravenous antibiotic treatment within 4 weeks before screening or oral antibiotic treatment within 2 weeks before screening;
11. Subjects who have received live vaccines/attenuated vaccines within 4 weeks before the screening visit or are known to receive live vaccines/attenuated vaccines during the 12-week treatment observation period;
12. Subjects who have used or plan to use lymphocyte-depleting agents/therapies, alkylating agents, total lymphoid irradiation, or other treatment methods during the study period;
13. Individuals who have previously received IL-6 and IL-6R inhibitor treatment;
14. Use of biological disease-modifying anti-rheumatic drugs (bDMARDs) within 4 weeks or 5 half-lives (whichever is longer) before randomization: such as TNF-α inhibitors, biosimilars, and RA drugs used in clinical trials;
15. Use of non-biological DMARDs other than MTX within 28 days before dosing (excluding chloroquine and hydroxychloroquine, subjects who have used leflunomide within 140 days before dosing or have undergone standard cholestyramine treatment or activated charcoal washout within 28 days before dosing are not eligible for the trial);
16. Receipt of intra-articular or extra-articular (intramuscular, intravenous) corticosteroid treatment within 28 days before dosing;
17. Participation in other drug clinical studies within 1 month or 5 half-lives (whichever is longer) of other trial drugs before screening;
18. Hepatitis B surface antigen (HBsAg) positive, or if hepatitis B core antibody (HBcAb) is positive, then HBV DNA is additionally checked and HBV DNA > lower limit of detection;
19. Screening period laboratory test values (only one retest is allowed) meet any of the following conditions:

    * Serum creatinine: Female subjects with serum creatinine > 1.4 mg/dL (124 μmol/L); male subjects with serum creatinine > 1.6 mg/dL (141 μmol/L);
    * ALT or AST > 1.5 times the upper limit of normal (ULN);
    * Platelet count < 80×10^9/L;
    * WBC < 3.0×10^9/L;
    * Total bilirubin > 1.5 times ULN;
    * Neutrophil count < 1.5×10^9/L;
    * Lymphocyte count < 0.5×10^9/L.
20. Pregnant or breastfeeding women, or female subjects with positive pregnancy tests during the screening period/baseline period, or subjects (including male subjects and their female spouses) who cannot take effective contraceptive measures from the screening period to 6 months after completion or termination of the trial;
21. Subjects whom the investigator deems otherwise unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving ACR50 at week 24 (W24). | 24 weeks
  Proportion of patients who achieving American College of Rheumatology 50% improvement criteria (ACR20) at week 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes